CLINICAL TRIAL: NCT04025593
Title: A Randomized, Phase 2 Study of Biomarker Guided Treatment in DLBCL
Brief Title: Biomarker Guided Treatment in DLBCL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, Deputy director of hematology department, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Guidance-01
Record Dates: First submitted 2019-07-17; First posted 2019-07-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Cyclophosphamide; Rituximab; Doxorubicin; Vincristine; Prednisone; ibrutinib; Lenalidomide; N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; Decitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RCHOP (Active Comparator)
  Interventions: Drug: Cyclophosphamide; Drug: Rituximab; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone
- RCHOPX (Experimental)
  Interventions: Drug: Cyclophosphamide; Drug: Rituximab; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone; Drug: Ibrutinib; Drug: Lenalidomide; Drug: chidamide; Drug: decitabine

INTERVENTIONS:
Drug: Cyclophosphamide — 750mg/m2 day 1
Drug: Rituximab — 375mg/m2 day 0
Drug: Doxorubicin — 50mg/m2 day 1
Drug: Vincristine — 1.4mg/m2, max 2mg day 1
Drug: Prednisone — 60mg/m2, max 100mg day 1-5
Drug: Ibrutinib — 420mg/day qd
  Arms: RCHOPX
Drug: Lenalidomide — 25mg day1-10
  Arms: RCHOPX
Drug: chidamide — 20mg day 1,4,8,11
  Arms: RCHOPX
Drug: decitabine — decitabine 10mg/m2 day-5 to day-1
  Arms: RCHOPX

SUMMARY:
This study is to investigate the strategy of biomarker guided treatment in diffuse large B cell lymphoma

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed diffuse large B-cell lymphoma, CD20 positive
* ECOG 0,1,2
* Life expectancy>6 months
* Informed consented
* IPI>1

Exclusion Criteria:

* Chemotherapy before
* Stem cell transplantation before
* History of malignancy except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix
* Uncontrollable cardio-cerebral vascular, coagulative, autoimmune, serious infectious disease
* Primary CNS lymphoma
* LVEF≤50%
* Lab at enrollment (Unless caused by lymphoma) Neutrophile<1.5*10^9/L Platelet<75*10^9/L ALT or AST >2*ULN,AKP or bilirubin >1.5*ULN Creatinine>1.5*ULN Other uncontrollable medical condition that may that may interfere the participation of the study Not able to comply to the protocol for mental or other unknown reasons Pregnant or lactation HIV infection If HbsAg positive, should check HBV DNA, DNA positive patients cannot be enrolled. If HBsAg negative but HBcAb positive (whatever HBsAb status), should check HBV DNA,DNA positive patients cannot be enrolled.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2019-07-17 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
complete response rate | 21 days after 6 cycles of treatment (each cycle is 21 days)

SECONDARY OUTCOMES:
progression free survival | 2 year
overall survival | 2 year
overall response rate | 21 days after 6 cycles of treatment (each cycle is 21 days)
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0 | Up to 30 days after completion of study treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No